CLINICAL TRIAL: NCT02192632
Title: Dermatologists' Educational Demonstration for Epiduo Application
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Dae Hun Suh, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ADP-BPO; 1402-051-555 (Registry Identifier: 1402-051-555)
Record Dates: First submitted 2014-07-14; First posted 2014-07-17 (Estimated); Last update posted 2015-03-17 (Estimated); Status verified 2015-03

CONDITIONS: Facial Acne; Local Adverse Effects

STUDY DESIGN:
Who Masked: Investigator

ARMS (3):
- Epiduo- dermatologist's detailed instruction (Experimental): After randomly assigned to side of epiduo application, half of total patients were also re-assigned into detailed instruction for application of epiduo from dermatologist
  Interventions: Drug: Epiduo once daily with detailed instruction for how to apply it
- Epiduo- drug insert only gruop (Experimental): After randomly assigned to side of epiduo application, half of total patients were also re-assigned into drug insert only group
  Interventions: Drug: Epiduo- once daily, simple instruction for application
- BPO group (Placebo Comparator): After randomly assigned to side of BPO application, patients apply BPO during 12 week
  Interventions: Drug: BPO once daily

INTERVENTIONS:
Drug: Epiduo once daily with detailed instruction for how to apply it
  Arms: Epiduo- dermatologist's detailed instruction
Drug: Epiduo- once daily, simple instruction for application
  Arms: Epiduo- drug insert only gruop
Drug: BPO once daily
  Arms: BPO group

SUMMARY:
The purpose of this study is to evaluate the efficacy and tolerability of this combination gel compared with BPO monotherapy in Korean patients, and test clinical practicability of dermatologists' educational demonstration for how to apply this gel in reducing uncomfortable irritations.

ELIGIBILITY:
Inclusion Criteria:

* mild to moderate acne were evaluated by Leeds revised acne grade from 2 to 6
* age: 18-40

Exclusion Criteria:

* pregnancy
* mental illness
* intake of oral isotretinoin within 6 months
* application of the other oral or topical acne medications
* chemical peeling or light based treatments within 6 weeks.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 85 (Actual)
Dates: Start 2014-01; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Percentile reduction of non-inflammatory & inflammatory acne lesions | 12 weeks
  Measurement of decreases in both non-inflammatory & inflammatory acne lesions

SECONDARY OUTCOMES:
Total number of local irriation effect counts (erythema, scaling, dryness, itching) | 12 week
  Calcuation of total number of local irriation effect counts (erythema, scaling, dryness, itching)

CONTACTS AND LOCATIONS:
Locations (1):
- Dermatology, Seoul National University, Seoul, Joungro, South Korea